CLINICAL TRIAL: NCT01933191
Title: A Randomised Placebo Controlled Cross-over Trial on Exercise Treatment of Dental Anxiety
Brief Title: Exercise Treatment of Dental Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Prof. Dr. Andreas Ströhle, Prof. Dr., Charite University, Berlin, Germany
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 221014
Record Dates: First submitted 2013-07-26; First posted 2013-09-02 (Estimated); Last update posted 2015-02-09 (Estimated); Status verified 2015-02

CONDITIONS: Dental Anxiety
Keywords: Dental Anxiety, Physical Activity, Dental Phobia; Cortisol, Amylase
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- physical acticity (Experimental): Experimental: Aerobic treadmill exercise (30 minutes, 70% VO2max)
  Interventions: Behavioral: Aerobic treadmill exercise; Behavioral: placebo exercise
- placebo exercise (Placebo Comparator): Aerobic treadmill exercise (30 minutes, 20% VO2max)
  Interventions: Behavioral: Aerobic treadmill exercise; Behavioral: placebo exercise

INTERVENTIONS:
Behavioral: Aerobic treadmill exercise — Experimental training: Aerobic treadmill exercise (30 minutes, 70% VO2max) prior to an elective minor dental procedures (e.g., extractions, endodontics, apicoectomies, dental restorations, periodontal treatment, dental implants).
  Other Names: physical activity VO2-70%
Behavioral: placebo exercise — placebo exercise: Aerobic treadmill exercise (30 minutes, 20% VO2max) prior to an elective minor dental procedures (e.g., extractions, endodontics, apicoectomies, dental restorations, periodontal treatment, dental implants).
  Other Names: physical activity VO2-20%

SUMMARY:
A single bout of physical activity (treadmill)immediately prior to the dental examination reduces anxiety in patients with dental phobia.

DETAILED DESCRIPTION:
The primary objective of the trial is to assess the anxiolytic efficacy of 30 minutes aerobic treadmill exercise versus placebo exercise in subjects experiencing high anxiety prior to a minor dental dental procedure.

Primary efficacy endpoint:

Change in the visual analogue scale (VAS) for anxiety before and after the intervention prior to the elective minor dental procedure

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients 18 years of age or older
* A total score of 12 points or more on the Dental Anxiety Scale at screening and baseline evaluations
* Scheduled appointment for an elective minor dental procedure
* Informed consent

Exclusion Criteria:

* Pregnant or lactating women
* Current diagnosis of any other DSM-IV, with the exception of other phobic disorders, social anxiety disorder or dysthymia
* Serious medical disorders which put subjects at risk if they have to exercise 30 minutes at 70% VO2max

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-08; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in VAS - visual analog scale | Baseline and one hour after dental intervention
  Change in the visual analogue scale (VAS) for anxiety

SECONDARY OUTCOMES:
Change from Baseline in cortisol level | Baseline and one hour
  Cortisol is one of the main hormones released by the body as a reaction to stress.
Change from Baseline in alpha-Amylase | Baseline and one hour after dental intervention
  Salivary alpha-Amylase

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Ströhle, Prof. Dr., Principal Investigator — Department of Psychiatry and Psychotherapie, CCM, Charité-Universitätsmedizin Berlin
Locations (1):
- Department of Psychiatry and Psychotherapy Campus Charité Mitte, Berlin, Germany